CLINICAL TRIAL: NCT00215358
Title: Study in Patients With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Director, Clinical Affairs, Dey
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DL-048
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2008-02

CONDITIONS: Asthma
Keywords: Asthma; Formoterol; Fumarate; Foradil
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate

INTERVENTIONS:
Drug: Formoterol Fumarate

SUMMARY:
The purpose of this study is to determine which dose of the investigational drug is safest and most effective compared to the control drug.

ELIGIBILITY:
Inclusion Criteria:

-Require regular use of an inhaled Beta-2-selective adrenergic agent

Exclusion Criteria:

* Active acute or chronic disorders of the respiratory system within one month prior to screening
* Smoking history within the past 12 months or greater than a lifetime 10 pack-year smoking history
* Recent surgical interventions such as lung lobectomy or resection (< one year), or cardiothoracic interventions
* Life-threatening systemic and debilitating diseases.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32
Dates: Start 2002-07; Primary Completion 2002-10 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Measure of lung function.

SECONDARY OUTCOMES:
Change in lung function, vital signs, physical examinations, clinical laboratory assessments, and adverse event reporting.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Denver, Colorado
  - Research Site, Medford, Oregon